

# TRIAL STATISTICAL ANALYSIS PLAN

c21342784-01

| | 48.60.8 |
|---|---|
| BI Trial No.: | 1368.3 |
| Title: | Safety, tolerability, and pharmacokinetics of two dose strengths of a single subcutaneous dose of BI 655130 and one single intravenous dose of BI 655130 in healthy male and female subjects (open-label, parallel group design). |
| Investigational<br>Product: | BI 655130 |
| Responsible trial statisticians: | |
| | Phone:<br>Fax: |
| | Phone: Fax: |
| Date of statistical analysis plan: | 06 FEB 2018 SIGNED |
| Version: | Final |

**Proprietary confidential information** 

© 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1368.3 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. TABLE OF CONTENTS

| TITLE | PAGE | 1 |
|--------------|------------------------------------------------|----|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | F TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| 5. | ENDPOINTS | |
| 5.1 | PRIMARY ENDPOINTS | |
| 5.2 | SECONDARY ENDPOINT | |
| <b>5.2.1</b> | Key secondary endpoint | |
| 5.2.2 | Secondary endpoint | |
| 5.3 | FURTHER ENDPOINTS | |
| 5.3.2 | Safety parameters | |
| 5.4 | OTHER VARIABLES | |
| 5.4.1 | Demographic and other baseline characteristics | |
| 5.4.2 | Treatment compliance and treatment exposure | 10 |
| <b>6.</b> | GENERAL ANALYSIS DEFINITIONS | |
| 6.1 | TREATMENTS | |
| <b>6.2</b> | IMPORTANT PROTOCOL VIOLATIONS | |
| 6.3 | SUBJECT SETS ANALYSED | |
| 6.4 | SUBGROUPS | |
| 6.5 | POOLING OF CENTRES | |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | PLANNED ANALYSIS | |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4 | PRIMARY ENDPOINTS | |
| 7.5 | SECONDARY ENDPOINT | |
| 7.5.1 | Key secondary endpoint | |
| 7.5.2 | Secondary endpoint | |
| 7.7 | EXTENT OF EXPOSURE | |
| <b>7.8</b> | SAFETY ANALYSIS | |
| 7.8.1 | Adverse events | 18 |

# **Boehringer Ingelheim**

| TSAP | ' for | ΒI | Trial | No: | 1368.3 |
|------|-------|----|-------|-----|--------|
|------|-------|----|-------|-----|--------|

| Page | 3 | of | 24 |
|------|---|----|----|

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Laboratory data ......20 7.8.2 7.8.3 **7.8.4** 7.8.5 Others 20 **7.8.6** Local tolerability .......21 8. REFERENCES. 22 \_\_\_\_\_23 HISTORY TABLE 24 **10.** 

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1368.3 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 | Flow chart of analysis phases for statistical analyses of AEs, safety | |
|---|---|---|
| | laboratory data and vital signs | 11 |
| Table 6.2: 1 | Important protocol violations | 12 |
| Table 6.3: 1 | Subject sets analysed | 13 |
| | History table | |

TSAP for BI Trial No: 1368.3 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

| Term | Definition / description |
|---|---|
| ADPC | Proper name of the analysis dataset containing PK concentrations per time-point or per time-interval |
| ADPP | Proper name of the analysis dataset containing calculated PK parameters |
| ADS | Analysis dataset |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| ANOVA | Analysis of variance |
| AST | Aspartate aminotransferase |
| $AUC_{0-\infty}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity |
| AUC0-tz | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| BI | Boehringer Ingelheim |
| BLQ | Below the lower limit of quantification |
| BMI | Body mass index |
| CARE | Clinical data analysis and reporting environment |
| CI | Confidence interval |
| Cmax | Maximum measured concentration of the analyte in plasma |
| CRF | Case Report Form |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic coefficient of variation |
| DBLM | Database lock meeting |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| ER | Exploratory reference treatment |
| EudraCT | European union drug regulating authorities clinical trials |
| gCV | Geometric coefficient of variation |

TSAP for BI Trial No: 1368.3 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|--------|----------------------------------------------|
| gMean | Geometric mean |
| ICH | International Conference On Harmonisation |
| IPV | Important protocol violation |
| MedDRA | Medical Dictionary For Regulatory Activities |
| NOA | Not analysed |
| NOR | No valid result |
| NOS | No sample available |
| on-trt | on-treatment |
| PK | Pharmacokinetics |
| PKS | Pharmacokinetic parameter analysis set |
| PV | Protocol Violation |
| Q1 | Lower Quartile |
| Q3 | Upper Quartile |
| R | Reference treatment |
| RAGe | Report appendix generator |
| RPM | Report Planning Meeting |
| SAE | Serious adverse event |
| SD | Standard Deviation |
| SDL | Subject data listing |
| SOC | System Organ Class |
| T | Test treatment |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper limit of normal range |

# 3. INTRODUCTION

As per ICH E9  $(\underline{1})$ , the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the CTP, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the CTP. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data will be stored in a trial database within the Oracle Clinical<sup>TM</sup> system.

The statistical analyses will be performed within the validated working environment CARE, including SAS<sup>TM</sup> (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SAS<sup>TM</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

PK parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version 6.3, Certara USA Inc., Princeton, NJ, USA).

TSAP for BI Trial No: 1368.3 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses described in this TSAP are in accordance with the statistical methods described in the CTP.

# 5. ENDPOINTS

# 5.1 PRIMARY ENDPOINTS

Primary endpoints are PK endpoints as defined in Section 5.5.1.1 of the CTP:

- $AUC_{0-tz}$  (area under the concentration-time curve of BI 655130 in plasma over the time interval from 0 to the last quantifiable data point)
- $C_{max}$  (maximum measured concentration of BI 655130 in plasma)

# 5.2 SECONDARY ENDPOINT

# 5.2.1 Key secondary endpoint

Not applicable.

# 5.2.2 Secondary endpoint

Secondary endpoint is  $AUC_{0-\infty}$  (area under the concentration-time curve of BI 655130 in plasma over the time interval from 0 extrapolated to infinity).

# 5.3 FURTHER ENDPOINTS

# **5.3.2** Safety parameters

#### CTP:

Safety and tolerability of the investigational drug will be assessed based on:

- Adverse events (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG
- Continuous ECG monitoring
- Vital signs (blood pressure, pulse rate)
- Local tolerability
- Oral body temperature

Local tolerability will be assessed as absence or presence of "swelling", "induration", "heat", "redness", "pain", or "other findings".

# 5.4 OTHER VARIABLES

# 5.4.1 Demographic and other baseline characteristics

**CTP**: At screening, the medical examination will include demographics including height and body weight, smoking and alcohol history, relevant medical history and concomitant therapy [...].

Age [years] will be determined as the difference between year of birth and year of informed consent.

BMI will be calculated as weight  $[kg] / (0.01 * height [cm])^2$ .

# 5.4.2 Treatment compliance and treatment exposure

Treatment compliance will not be analysed as a specific endpoint, cf. Section 4.3 of the CTP.

Treatment exposure is defined as the total dose of BI 655130 per subject.

Additionally, the duration of infusion per subject is calculated for the treatment group of subjects who receive BI 655130 intravenously.

# 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

or

For basic study information on treatments to be administered, assignments of dose groups, and selection of doses, cf. Section 4 of the CTP.

Subjects were planned to be treated either with one single dose of

- as subcutaneous (SC) injection (exploratory reference treatment (ER))
  - or
    as intravenous (IV) infusion (reference treatment (R))
- as SC injection (test treatment (T)).

For statistical analysis of AEs, safety laboratory data and vital signs, the following analysis phases are defined for each subject:

Table 6.1: 1 Flow chart of analysis phases for statistical analyses of AEs, safety laboratory data and vital signs

| Study analysis phase | Label | Start (inclusive) | End (exclusive) |
|---|---|---|---|
| Screening | Screening | Date of informed consent | Date/time of administration of study drug |
| On-treatment | BI SC, or<br>BI IV or<br>BI SC,<br>respectively | Date/time of administration of study drug | 0:00 AM on day after<br>subject's trial termination<br>date |

CTR Section 15, Appendix 16.1.9.2.8.2 and Appendix 16.1.9.2.8.3 AE displays will present results for the on-treatment phase only.

In CTR Section 15 AE tables (but not in Appendix 16.1.9.2.8.2 and Appendix 16.1.9.2.8.3 AE tables), the following total will be provided in addition:

• "Total on-trt BI", defined as the total over all on-treatment phases involving BI 655130 CTR Appendix 16.1.9.2.8.1 displays will present results for the screening and on-treatment phases.

Additionally to the totals defined above, the following total will be provided in CTR Section 16.1.9.2.8.1 AE tables:

• "Total", defined as the total over all study phases (incl. screening and on-treatment).

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

# 6.2 IMPORTANT PROTOCOL VIOLATIONS

Consistency check listings (for identification of violations of time windows) and a list of protocol deviations (e.g. deviations in drug administration) will be provided to be discussed at the RPM/DBLM. At this meeting, each protocol deviation must be assessed to determine whether it is an IPV. For definition of IPVs, and for the process of identification of these, refer to the BI reference document "Protocol Violation Handling Definitions" (2).

If any IPVs are identified, they are to be summarised into categories and will be captured in the RPM/DBLM minutes via an accompanying Excel spreadsheet (3). The following table contains the categories which are considered to be IPVs in this trial. If the data show other IPVs, this table will be supplemented accordingly by the time of the RPM/DBLM.

IPVs will be summarised and listed.

Table 6.2: 1 Important protocol violations

| Category Description / Code | | Description |
|---|---|---|
| A | | Entrance criteria not met |
| | A1 | Inclusion criteria violated |
| | A2 | Exclusion criteria violated |
| В | | Informed consent |
| | B1 | Informed consent not available |
| | B2 | Informed consent too late |
| C | | Trial medication and randomisation |
| | C1 | Incorrect trial medication taken |
| | C3 | Non-compliance |
| | C5 | Incorrect intake of trial medication |
| D | | Concomitant medication |
| | D1 | Concomitant medication with the potential to affect the assessment of the trial medication |
| E | | Missing data |
| | | None <sup>1</sup> |
| G | | Other trial specific important violations |
| | G1 | Certain violations of procedures used to measure primary PK data |

Violations C1, C2, C5 and G1 can only be detected at the trial site.

Source: BI reference document "Protocol Violation Handling Definitions" [001-MCS-50-413\_RD-01] (2).

<sup>&</sup>lt;sup>1</sup> Missing visits, evaluations, and tests will be considered missing data, not PVs

# 6.3 SUBJECT SETS ANALYSED

The following subject sets will be defined for statistical analysis:

- Treated set (TS):
  This subject set includes all subjects who received study drug.
- Pharmacokinetic parameter set (PKS):
   This subject set includes all subjects of the TS who provide at least one observation for at least one primary or secondary PK endpoint without important PVs with respect to the statistical evaluation of PK endpoints, as defined in Section 7.3.1 and Section 7.3.2 of the CTP.

The discussion of all exceptional cases and problems and the decisions on the allocation of subjects to analysis sets will be made at latest at the RPM/DBLM.

Table 6.3: 1 Subject sets analysed

| | Subject set | |
|--------------------------------|-------------|-----|
| Class of endpoint | TS | PKS |
| Disposition | X | |
| Exposure | X | |
| IPVs | X | |
| Demographic/baseline endpoints | X | |
| Other safety parameters | X | |
| PK endpoints | | X |

# 6.4 SUBGROUPS

A subgroup analysis is not planned.

# 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

# 6.6 HANDLING OF MISSING DATA AND OUTLIERS

CTP: If a subject is removed from or withdraws from the trial prior to first administration of trial medication, the data of this subject will not be entered in the case report form (CRF) or trial database and will not be reported in the clinical trial report (CTR). If a subject is removed from or withdraws from the trial after first administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF. In this case, the data will be included in the CRF/trial database and will be reported in the CTR.

**CTP**: With respect to safety evaluations, it is not planned to impute missing values.

The only exceptions where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards (see 001-MCG-156 RD-01 (4)).

Missing data and outliers of PK data are handled according to BI standards (see 001-MCS-36-472\_RD-01) (5). **CTP**: Drug concentration data identified with NOS (no sample available), NOR (no valid result), NOA (not analysed), BLQ (below the lower limit of quantification), or NOP (no peak detectable) will be displayed as such and not replaced by zero at any time point (this rule also applies also to the lag phase, including the predose values).

**CTP**: For the non-compartmental analysis, concentration data identified with NOS, NOR or NOA will generally not be considered. Concentration values in the lag phase identified as BLQ or NOP will be set to zero. All other BLQ/NOP values of the profile will be ignored. The lag phase is defined as the period between time zero and the first time point with a concentration above the quantification limit.

# 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

For safety measurements baseline is defined as the last measurement before study drug administration.

Time windows are defined in Section 6.1 of the CTP. Adherence to time windows will be checked at the RPM/DBLM.

# 7. PLANNED ANALYSIS

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries" (001-MCG-159) (10).

The individual values of all subjects will be listed. Listings will generally be sorted by treatment group, subject number and visit (if visit is applicable in the respective listing). AE listings will be sorted by assigned analysis phase (see <u>Table 6.1: 1</u> for a definition of analysis phases). The listings will be contained in Appendix 16.2 (SDL) of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For plasma concentrations as well as for all PK parameters, the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

The data format for descriptive statistics of plasma concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment. Percentages will be rounded to one decimal place. The category missing will be displayed if and only if there actually are missing values. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not.

# 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR.

# 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases will be coded according to the most recent version of MedDRA. Concomitant medication will be coded according to the most recent version of the World Health Organisation – Drug Dictionary.

Only descriptive statistics are planned for this section of the CTR.

A medication will be considered concomitant to a treatment, if it

- is ongoing at the time of administration of the respective treatment or
- starts within the analysis phase of the respective treatment (see <u>Section 6.1</u> for a definition of treatments and analysis phases).

# 7.3 TREATMENT COMPLIANCE

Treatment compliance will not be analysed as a specific endpoint, but will be assessed for the treatment group receiving BI 655130 intravenously based on the duration of infusions (descriptive statistics of duration) and dose per infusion (descriptive statistics of the administered dose per infusion). Any deviations from complete intake will be addressed in the RPM/DBLM (cf. Section 6.2) and described in the CTR.

# 7.4 PRIMARY ENDPOINTS

Analysis of relative BA of primary endpoints  $AUC_{0-tz}$  and  $C_{max}$  of BI 655130 in plasma will be performed as defined in Sections 7.1.3 and 7.3.1 of the CTP.

The statistical model for the primary analysis (comparison of subcutaneous versus intravenous administration of of BI 655130) is an ANOVA model on the logarithmic scale including an effect for "treatment group" as defined in Sections 7.1.3 and 7.3.1 of the CTP.

Primary PK endpoints will also be assessed descriptively. The analysis of standard PK parameters is performed according to BI standards (5) [001-MCS-36-472\_RD-01].

# Exclusion of PK parameters

The ADS ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS are based on PK parameter values which are not flagged for exclusion, i.e. with APEXC equal to "Included".

# Exclusion of plasma concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to "ALL CALC", the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to "DESC STATS" the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition "TIME VIOLATION" or "TIME DEVIATION", the value can be used for further analyses based on actual times. If ACEXCO is set to "HALF LIFE", the value will be excluded from half-life calculation only; the value is included for all other analyses.

Further details are given in 001-MCS-36-472\_RD-01 "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (5) and 001-MCS-36-472\_RD-03 "Description of Analytical Transfer Files and PK/PD Data Files" (6).

# 7.5 SECONDARY ENDPOINT

# 7.5.1 Key secondary endpoint

Not applicable.

# 7.5.2 Secondary endpoint

The secondary PK endpoint  $AUC_{0-\infty}$  will be analysed in the same way as described for the primary PK endpoint.

Descriptive analyses of the secondary PK endpoint will be performed according to BI standards (5) [001-MCS-36-472\_RD-01].

See <u>Section 7.4</u> of this TSAP for details regarding exclusion of PK parameters and plasma concentrations.

# 7.7 EXTENT OF EXPOSURE

Only descriptive statistics are planned for this section of the CTR, see also <u>Section 7.3</u>.

# 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

# 7.8.1 Adverse events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs.

For analysis, multiple AE occurrence data on the eCRF will be collapsed into one event provided that all of the following applies:

- All AE attributes are identical (lower level term, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AESI)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started at most 1 hour after the first occurrence ended)

For further details on summarization of AE data, please refer to "Analysis and Presentation of Adverse Event Data from Clinical Trial" (7) [001-MCG-156] and "Handling of missing and incomplete AE dates" (4) [001-MCG-156\_RD-01].

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to the screening phase or on-treatment phase as defined in Section 6.1.

An overall summary of AEs will be presented. This overall summary will comprise summary statistics for the class of other significant AEs according to ICH E3 and for the class of AESIs.

**CTP:** The AESI in this trial is hepatic injury, as defined by the following alterations of hepatic laboratory parameters:

- an elevation of AST and/or  $ALT \ge 3$ -fold ULN combined with an elevation of total bilirubin  $\ge 2$ -fold ULN measured in the same blood sample, and/or
- aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

According to ICH E3 (9), AEs classified as "other significant" need to be reported and will include those non-serious and non-significant AEs

- (i) which are marked haematological or other lab abnormalities, or
- (ii) which were reported with "action taken = discontinuation" or "action taken = reduced", or (iii) which lead to significant concomitant therapy as identified by the Clinical

Monitor/Investigator at a Medical Quality Review Meeting.

The frequency of subjects with AEs will be summarised by treatment, primary SOC and preferred term. AEs which were considered by the investigator to be drug related will be summarised separately. Separate tables will also be provided for subjects with SAEs, subjects with AESIs and subjects with other significant AEs (according to ICH E3 (9)). The frequency of subjects with AEs and the frequency of subjects with AEs considered by the investigator to be drug related will also be summarised by maximum intensity, primary SOC and preferred term.

The SOCs and preferred terms within SOCs will be sorted by descending frequency overall treatment groups.

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised by treatment, primary SOC and preferred term. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarised.

# 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards (8). If possible, analyses will be based on original values. If multiple reference ranges apply for a parameter (e.g. due to different age groups), analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range.

Descriptive statistics of laboratory values over time and for the difference from baseline (see <u>Section 6.7</u>) will be provided. Frequency tables of changes between baseline and last value on treatment with respect to the reference range will be presented.

Possibly clinically significant abnormal laboratory values are only those identified either in the Investigator's comments or at the RPM/DBLM at the latest. It is the Investigator's responsibility to decide whether a lab value is clinically significant abnormal or not. Standard or project-specific rules for flagging clinically significant values in an automated manner will not be applied in this study.

Clinically relevant findings in laboratory data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

# 7.8.3 Vital signs

The analyses of vital signs (blood pressure, pulse rate, body temperature) will be descriptive in nature. Descriptive statistics of vital signs over time and for the difference from baseline (see Section 6.7) will be provided.

Body weight will only be listed.

Clinically relevant findings in vital signs data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

# 7.8.4 ECG

Abnormal findings in ECG will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such. No separate listing or analysis of ECG data will be prepared.

# **7.8.5** Others

Physical examination findings will be reported as relevant medical history/baseline condition (i.e., a condition already existent before intake of study drug) or as AE and will be summarised as such. No separate listing or analysis of physical examination will be prepared.

Matching pairs for subjects included in the BI SC and BI IV treatment group will be summarized in a table and a listing displaying the matching criteria.

# 7.8.6 Local tolerability

Local tolerability (absence or presence of "swelling", "induration", "heat", "redness", "pain", or "other findings") will be summarized with counts and percentages overall (i.e. over all time points) as well as by time point.

# 8. REFERENCES

1 *CPMP/ICH/363/96:* "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version.

9 *CPMP/ICH/137/95*: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version

TSAP for BI Trial No: 1368.3 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1368.3 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **10. HISTORY TABLE**

History table Table 10: 1

| Version | Date<br>(DD-MMM-<br>YY) | Author | | Sections changed | Brief description of change |
|---|---|---|---|---|---|
| Final | 06-FEB-18 | | | None | This is the final TSAP without any modification |
| | | ( | ), | | |
| | | ( | ) | | |